CLINICAL TRIAL: NCT04313595
Title: A Wearable Device for Breathing Frequency Monitoring: a Pilot Study on Patients With Muscular Dystrophy
Brief Title: Device for Breathing Frequency Monitoring in Muscular Dystrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 534
Record Dates: First submitted 2020-02-26; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Muscular Dystrophies
MeSH Terms: conditions — Muscular Dystrophies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breathing frequency monitoring (Experimental)
  Interventions: Device: RespirHó

INTERVENTIONS:
Device: RespirHó — The system is a wearable, unobtrusive inertial-sensor-based device for long-term breathing pattern monitoring, also during daily life activities. It consists of three IMU-sensor units (3-axis accelerometer, 3-axis gyroscope, 3-axis magnetometer), positioned respectively on the patient's abdomen and thorax, and on a body area integral with thorax but not affected by espiratory movements. The peripheral units, placed on thorax and abdomen are used to record orientation changes during respiratory movements. The third unit is a central reference unit (hereafter CRU) that receives data from the other two units, save them on an SD card and communicate via Bluetooth with a smartphone / tablet / PC. Moreover, this unit detects only non-respiratory movement, representing not only a pure source of "noise" that must be removed from the thoracic and bdominal signals, but also a pure source of additional information regarding the state of ctivity of the subject .

SUMMARY:
Patients at risk of developing respiratory dysfunctions, such as patients with severe forms of muscular dystrophy, need a careful respiratory assessment, and periodic follow-up visits to monitor the progression of the disease. Continuous monitoring of respiratory activity pattern at home could give additional understandings about disease progression, flanking traditional, intermittent, cardiopulmonary evaluations, allowing prompt clinical intervention, and anticipating respiratory dysfunction. The main objective of the present study is thus to investigate the feasibility of using an innovative wearable device for respiratory monitoring, especially breathing frequency variation assessment, in patients with muscular dystrophy. The comparison between the measurements of breathing frequency obtained by using the IMU-based device and by using the reference method provided optimal results, in terms of accuracy errors, correlation and agreement. Participants positively evaluated the device for what concerns ease of use, comfort, usability and wearability. Moreover, preliminary results confirmed that breathing frequency is an interesting breathing parameter to monitor, at the clinic and at home, because it strongly correlates with the main indexes of respiratory function

ELIGIBILITY:
Inclusion criteria:

* documented DMD or LGMD2
* loss of independent ambulation (wheelchair-bound patients)
* ability to understand and follow test instructions and to report pain and discomfort.

Exclusion criteria:

* presence of metal implants and cardiac pacemakers
* relevant concomitant comorbidities (e.g.epilepsy)
* behaviour and/or psychiatric disorders (e.g. emotional problems, anxiety, panic attacks).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-07-29 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Safety of the device | After 24 hours of continued use
  Recording of any adverse events
Usability of the device (System Usability Scale) | After 24 hours of continued use
  System Usability Scale (SUS acceptance and wearability of the device):the scores range from 0 to 100 in 2.5-point increments, with higher values meaning high perceived usability of the system
Acceptability of the device (Technological Acceptance Measure) | After 24 hours of continued use
  Technological Acceptance Measure (TAM) questionnaire appropriate for the medical device: with higher values meaning high acceptance of the system

SECONDARY OUTCOMES:
Accuracy in measuring the breathing frequency | Immediately after application of the device
  Comparison between the measures of respiratory rate by using the device and by using already validated instrumentation: Optoelectronic Plethysmography (OEP), optoelectronic movement analysis system.
  Chest wall movements during breathing are simultaneously recorded by the RespirHó device and by Optoelectronic Plethysmography (OEP), in static conditions, and in particular, in supine and seated positions.
  OEP allows assessment of ventilatory and breathing pattern by measuring chest-wall movements related to breathing, by using motion capture principles.
  Using OEP as reference method it is possible to compare the data recorded with the thoracic and abdominal units of the device RespirHó with those obtained by using OEP for the thoracic and abdominal compartments

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Medea, Bosisio Parini, Lecco, Italy

IPD SHARING:
Plan to Share IPD: No